CLINICAL TRIAL: NCT04639960
Title: Effects of Modulation of the Dopaminergic System Using Risperidone on Memory and Executive Processes in Individuals With 22q11.2 Deletion Syndrome
Brief Title: Neuroprotective Effects of Risperdal on Brain and Cognition in 22q11 Deletion Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruitment of participants and end of funding
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Stephan Eliez, Principal Investigator, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PB_201601540
Record Dates: First submitted 2020-11-03; First posted 2020-11-23 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: 22q11.2 Deletion Syndrome
MeSH Terms: conditions — DiGeorge Syndrome | interventions — Risperidone

STUDY DESIGN:
Intervention Model Description: double blind placebo design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the pharmacy has prepared the randomization. group membership will be revealed at the end of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Risperidone (Experimental)
  Interventions: Drug: Risperdal
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Risperdal — Twelve weeks of treatment with a gradual increase of dosage over one week and a gradual decrease over two weeks.
  Other Names: risperidone
  Arms: Risperidone
Drug: Placebo — Twelve weeks of placebo treatment.
  Arms: Placebo

SUMMARY:
Chromosome 22q11.2 deletion syndrome (22q11DS) is a neurogenetic condition associated with a high risk of psychiatric disorders, including schizophrenia spectrum disorders. This population is characterized by a particular neurocognitive profile and atypical brain development. Risperidone is a second-generation antipsychotic, inhibitor of dopaminergic receptors. Used in the treatment of psychosis, risperidone is frequently prescribed in 22q11DS, for example to treat a psychotic episode. Research on an animal model of 22q11DS (LgDel+/- mice) shows that administering an antipsychotic for 12 days during a critical period of brain development (adolescence) prevents deleterious neuronal changes and improves behavioral performance in mice. The aim of this study is therefore to replicate the results found in mice and to identify a long-term neuroprotective effect.

This study is inspired on the one hand by the families who share with us the difficulties of individuals affected by 22q11DS on a daily basis, but also by the encouraging results of studies conducted on mice.

DETAILED DESCRIPTION:
In a double-blind placebo design, this study investigates the effects of a 12 weeks treatment of risperidone (vs placebo) for participants with 22q11DS without psychotic symptoms.

The research hypothesis of this study is that a short-term (12 weeks) risperidone (Risperdal®) treatment during a critical phase of development (adolescence) will result in improved cognitive performance and brain changes observable using brain imaging techniques (Magnetic resonance Imaging, MRI and Electroencephalography, EEG). In addition, the beneficial effects will be observable in a follow-up evaluation, 6 months after the of treatment.

Risperdal® is a marketed product and is listed in the Swiss Compendium (2015). However, it is not used according to its indication for the treatment of psychotic disorders. The treatment will be administered orally in the form of capsules containing the ground tablet in order to preserve the double-blind procedure (meaning that neither the examiner nor the patient knows whether the capsule contains the active ingredient risperidone or a placebo). The dose will be individually adjusted according to the weight of each participant. The lowest dose recommended in the Swiss Compendium is 0.25 mg/day for children. Therefore this dos will be prescribe at the beginning of the treatment and then gradually increased to 0.25 mg gradually over 7 days. For individuals weighing less than 50 kg, the recommended dose is 0.5 mg/day, this dose will not be exceeded for these individuals. For individuals over 50 kg, the recommended dose is 1 mg/day. this dose will not exceeded for individuals over 50 kg. However, in order to adapt as closely as possible to the different weight categories, a dose of 0.75 mg will be given to the 51 to 70 kg weight category, and a maximum dose of 1 mg to individuals over 70 kg. Treatment will also be discontinued in progressive stages over a period of two weeks.

Each participant will complete a series of evaluations including cognitive tests and brain imaging (MRI and EEG) on 3 occasions: the 1st before the treatment period (baseline), the 2nd at the end of the treatment period (short-term effect) and the 3rd 6 months after the end of treatment (long-term effect).

ELIGIBILITY:
Inclusion Criteria:

* Male or female with confirmed 22q11DS diagnosis.
* Minimum age of 8 years or maximum age of 25 years and 11 months.
* Sufficient verbal expression and comprehension skills to understand and follow instructions based on initial interview.

Exclusion Criteria:

* Participants younger than 8 years and older that 25 years and 11 months.
* Previous adverse experience with risperidone
* Psychotic symptoms requiring sustained antipsychotic treatment
* Corrected QT (QTc) distance at baseline electrocardiogram above 460 milliseconds or elongation at control electrocardiogram (Day 6 of treatment) superior to 30 milliseconds with functional complaint.
* Pregnancy or breastfeeding.

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Conners' Continuous performance test, third edition (CPT-3) | CPT-3 pre-treatment
  Participants are instructed to press a button every time a letter appeared on the screen, except for the letter X where participants had to withhold their answer. Variables of interest are Detectability, Omission, Commission, Perseveration, Hit Reaction Time, Hit Reaction time Standard Deviation, Variability, Hit Reaction Time Block Change and Hit Reaction Time Inter- Stimulus Intervals Change.
Conners' Continuous performance test, third edition (CPT-3) | CPT-3 One week after treatment
  Participants are instructed to press a button every time a letter appeared on the screen, except for the letter X where participants had to withhold their answer. Variables of interest are Detectability, Omission, Commission, Perseveration, Hit Reaction Time, Hit Reaction time Standard Deviation, Variability, Hit Reaction Time Block Change and Hit Reaction Time Inter- Stimulus Intervals Change.
Conners' Continuous performance test, third edition (CPT-3) | CPT-3 six month after treatment
  Participants are instructed to press a button every time a letter appeared on the screen, except for the letter X where participants had to withhold their answer. Variables of interest are Detectability, Omission, Commission, Perseveration, Hit Reaction Time, Hit Reaction time Standard Deviation, Variability, Hit Reaction Time Block Change and Hit Reaction Time Inter- Stimulus Intervals Change.
Stroop Task | Stroop inhibition ratio pre-treatment
  To measure the cost of cognitive inhibition in time, an inhibition ratio score is computed by dividing the raw score from the Stroop condition (participants have to name the color of the ink even though the word spells a different color) by the raw score in the color naming condition (participants are instructed to name rectangles of colors as fast as possible). This score reflects the cognitive cost of inhibiting the reading process. A ratio value close to 1 indicates a lesser cost of inhibition.
Stroop Task | Stroop inhibition ratio one week after treatment
  To measure the cost of cognitive inhibition in time, an inhibition ratio score is computed by dividing the raw score from the Stroop condition (participants have to name the color of the ink even though the word spells a different color) by the raw score in the color naming condition (participants are instructed to name rectangles of colors as fast as possible). This score reflects the cognitive cost of inhibiting the reading process. A ratio value close to 1 indicates a lesser cost of inhibition.
Stroop Task | Stroop inhibition ratio six month after treatment
  To measure the cost of cognitive inhibition in time, an inhibition ratio score is computed by dividing the raw score from the Stroop condition (participants have to name the color of the ink even though the word spells a different color) by the raw score in the color naming condition (participants are instructed to name rectangles of colors as fast as possible). This score reflects the cognitive cost of inhibiting the reading process. A ratio value close to 1 indicates a lesser cost of inhibition.
Letter-number sequencing | Letter-number Sequencing pre-treatment
  A working memory subtest of the Wechsler Adult Intelligence Scale (WAIS) and the Wechsler Intelligence Scale for Children (WISC) in which the participant must sequence a random order of numbers and letters. Specifically, the participant must first say the numbers in ascending order and then the letters in alphabetical order. Longest sequence of letters and numbers correctly ordered
Letter-number sequencing | Letter-number Sequencing one week after treatment
  A working memory subtest of the Wechsler Adult Intelligence Scale (WAIS) and the Wechsler Intelligence Scale for Children (WISC) in which the participant must sequence a random order of numbers and letters. Specifically, the participant must first say the numbers in ascending order and then the letters in alphabetical order. Longest sequence of letters and numbers correctly ordered
Letter-number sequencing | Letter-number Sequencing six month after treatment
  A working memory subtest of the Wechsler Adult Intelligence Scale (WAIS) and the Wechsler Intelligence Scale for Children (WISC) in which the participant must sequence a random order of numbers and letters. Specifically, the participant must first say the numbers in ascending order and then the letters in alphabetical order. Longest sequence of letters and numbers correctly ordered
Color Trails test (CTT) | CTT flexibility ratio pre-treatment
  To measure the cost of task switching, a flexibility ratio was calculated to account for processing speed by dividing the time to complete part B (drawing a line between number following chronological order while alternating between colors) by time to complete part A (drawing a line between number following chronological order). Value closer to 1 indicate better flexibility.
Color Trails test (CTT) | CTT flexibility ratio one week after treatment
  To measure the cost of task switching, a flexibility ratio was calculated to account for processing speed by dividing the time to complete part B (drawing a line between number following chronological order while alternating between colors) by time to complete part A (drawing a line between number following chronological order). Value closer to 1 indicate better flexibility.
Color Trails test (CTT) | CTT flexibility ratio six month after treatment
  To measure the cost of task switching, a flexibility ratio was calculated to account for processing speed by dividing the time to complete part B (drawing a line between number following chronological order while alternating between colors) by time to complete part A (drawing a line between number following chronological order). Value closer to 1 indicate better flexibility.
Cambridge Neuropsychological Test Automated Battery (CANTAB) | CANTAB pre-treatment
  The Motor Screening test (MOT) is a training procedure designed screen for difficulties with vision, movement, or comprehension and ascertains that the subject can follow simple instructions, as well as familiarising them with the touch screen.
  Intra-Extra Dimensional Set Shift (IED) is a test of rule acquisition and reversal. It features visual discrimination and attentional set formation maintenance, shifting and flexibility of attention.
  Spatial Working Memory (SWM) is a test of the subject's ability to retain spatial information and to manipulate remembered items in working memory. It is a self-ordered task, which also assesses heuristic strategy.
  Stop Signal Task (SST) is a classic stop signal response inhibition test, which uses staircase functions to generate an estimate of stop signal reaction time. This test gives a measure of an individual's ability to inhibit a prepotent response.
Cambridge Neuropsychological Test Automated Battery (CANTAB) | CANTAB one week after treatment
  The Motor Screening test (MOT) is a training procedure designed screen for difficulties with vision, movement, or comprehension and ascertains that the subject can follow simple instructions, as well as familiarising them with the touch screen.
  Intra-Extra Dimensional Set Shift (IED) is a test of rule acquisition and reversal. It features visual discrimination and attentional set formation maintenance, shifting and flexibility of attention.
  Spatial Working Memory (SWM) is a test of the subject's ability to retain spatial information and to manipulate remembered items in working memory. It is a self-ordered task, which also assesses heuristic strategy.
  Stop Signal Task (SST) is a classic stop signal response inhibition test, which uses staircase functions to generate an estimate of stop signal reaction time. This test gives a measure of an individual's ability to inhibit a prepotent response.
Cambridge Neuropsychological Test Automated Battery (CANTAB) | CANTAB six month after treatment
  The Motor Screening test (MOT) is a training procedure designed screen for difficulties with vision, movement, or comprehension and ascertains that the subject can follow simple instructions, as well as familiarising them with the touch screen.
  Intra-Extra Dimensional Set Shift (IED) is a test of rule acquisition and reversal. It features visual discrimination and attentional set formation maintenance, shifting and flexibility of attention.
  Spatial Working Memory (SWM) is a test of the subject's ability to retain spatial information and to manipulate remembered items in working memory. It is a self-ordered task, which also assesses heuristic strategy.
  Stop Signal Task (SST) is a classic stop signal response inhibition test, which uses staircase functions to generate an estimate of stop signal reaction time. This test gives a measure of an individual's ability to inhibit a prepotent response.
15 signs & 15 words | 15 signs & 15 words pre-treatment
  15 signs & 15 words is a homemade episodic memory task inspired by the Rey Auditory Verbal Learning Test (Rey, 1958). Participants are required to learn 15 common French words and 15 signs (drawings made out of 1 or 2 basic geometrical forms). After delays of thirty minutes, one day, one week and one month, participants are asked to freely recall the words and the signs they remembered. They are also asked to recognize the target items form a list of distractors. Variables of interest are (1) learning score = Maximum number of items correctly recalled during learning divided by the number of trials to reach learning criterion. Low score indicates poor learning. (2) Retention % thirty minutes/on day/one week/one month = Number of items recalled after each delay in time divided by the maximum of items recalled during learning. Low score indicates poor memory.
15 signs & 15 words | 15 signs & 15 words on week after treatment
  15 signs & 15 words is a homemade episodic memory task inspired by the Rey Auditory Verbal Learning Test (Rey, 1958). Participants are required to learn 15 common French words and 15 signs (drawings made out of 1 or 2 basic geometrical forms). After delays of thirty minutes, one day, one week and one month, participants are asked to freely recall the words and the signs they remembered. They are also asked to recognize the target items form a list of distractors. Variables of interest are (1) learning score = Maximum number of items correctly recalled during learning divided by the number of trials to reach learning criterion. Low score indicates poor learning. (2) Retention % thirty minutes/on day/one week/one month = Number of items recalled after each delay in time divided by the maximum of items recalled during learning. Low score indicates poor memory.
15 signs & 15 words | 15 signs & 15 words six month after treatment
  15 signs & 15 words is a homemade episodic memory task inspired by the Rey Auditory Verbal Learning Test (Rey, 1958). Participants are required to learn 15 common French words and 15 signs (drawings made out of 1 or 2 basic geometrical forms). After delays of thirty minutes, one day, one week and one month, participants are asked to freely recall the words and the signs they remembered. They are also asked to recognize the target items form a list of distractors. Variables of interest are (1) learning score = Maximum number of items correctly recalled during learning divided by the number of trials to reach learning criterion. Low score indicates poor learning. (2) Retention % thirty minutes/on day/one week/one month = Number of items recalled after each delay in time divided by the maximum of items recalled during learning. Low score indicates poor memory.
Magnetic Resonance Imaging (MRI) T1-weighted | MRI T1-weighted pre-treatment
  T1 structural images are collected to obtain accurate measurements of regional developmental changes in cortical morphometry comprising estimates of cortical volume, thickness and surface area. An MPRAGE T1-weighted sequence is employed with the following parameters: TR = 2500 ms, TE = 3 ms, flip angle = 8°, matrix acquisition = 256 × 256, field of view = 23.5 cm, slice thickness = 3.2 mm, 192 slices.
Magnetic Resonance Imaging (MRI) T1-weighted | MRI T1-weighted one week after treatment
  T1 structural images are collected to obtain accurate measurements of regional developmental changes in cortical morphometry comprising estimates of cortical volume, thickness and surface area. An MPRAGE T1-weighted sequence is employed with the following parameters: TR = 2500 ms, TE = 3 ms, flip angle = 8°, matrix acquisition = 256 × 256, field of view = 23.5 cm, slice thickness = 3.2 mm, 192 slices.
Magnetic Resonance Imaging (MRI) T1-weighted | MRI T1-weighted six month after treatment
  T1 structural images are collected to obtain accurate measurements of regional developmental changes in cortical morphometry comprising estimates of cortical volume, thickness and surface area. An MPRAGE T1-weighted sequence is employed with the following parameters: TR = 2500 ms, TE = 3 ms, flip angle = 8°, matrix acquisition = 256 × 256, field of view = 23.5 cm, slice thickness = 3.2 mm, 192 slices.
MRI Spectroscopy | MRI Spectroscopy pre-treatment
  Acquisition of Single-voxel MRI Spectroscopy investigates changes in excitatory/inhibitory balance throughout development. More in detail, a Works-In-Progress (WIP) SVS (Single Voxel Spectroscopy) spin-echo sequence is used provided by Siemens and designed for detecting the GABA (Gamma-AminoButyric Acid) 1H MRS signal at 3 ppm in brain. 3 ROIs are selected: Anterior cingulate cortex (voxel size: 15 x 35 x 40, 98 avg), right hippocampus (voxel size: 20 x 30 x 40, 150 avg) and temporal cortex (voxel size: 30 x 30 x 30, 120 avg) that are manually placed during each session. Each sequence lasts around 7 minutes and patients are allowed to watch a video of their choice during the acquisition.
MRI Spectroscopy | MRI Spectroscopy one week after treatment
  Acquisition of Single-voxel MRI Spectroscopy investigates changes in excitatory/inhibitory balance throughout development. More in detail, a Works-In-Progress (WIP) SVS (Single Voxel Spectroscopy) spin-echo sequence is used provided by Siemens and designed for detecting the GABA (Gamma-AminoButyric Acid) 1H MRS signal at 3 ppm in brain. 3 ROIs are selected: Anterior cingulate cortex (voxel size: 15 x 35 x 40, 98 avg), right hippocampus (voxel size: 20 x 30 x 40, 150 avg) and temporal cortex (voxel size: 30 x 30 x 30, 120 avg) that are manually placed during each session. Each sequence lasts around 7 minutes and patients are allowed to watch a video of their choice during the acquisition.
MRI Spectroscopy | MRI Spectroscopy six month after treatment
  Acquisition of Single-voxel MRI Spectroscopy investigates changes in excitatory/inhibitory balance throughout development. More in detail, a Works-In-Progress (WIP) SVS (Single Voxel Spectroscopy) spin-echo sequence is used provided by Siemens and designed for detecting the GABA (Gamma-AminoButyric Acid) 1H MRS signal at 3 ppm in brain. 3 ROIs are selected: Anterior cingulate cortex (voxel size: 15 x 35 x 40, 98 avg), right hippocampus (voxel size: 20 x 30 x 40, 150 avg) and temporal cortex (voxel size: 30 x 30 x 30, 120 avg) that are manually placed during each session. Each sequence lasts around 7 minutes and patients are allowed to watch a video of their choice during the acquisition.
MRI Resting State | MRI resting state pre-treatment
  Functional MRI sequence without stimulation (resting-state fMRI) scans are employed to assess the longitudinal changes in regional activity and functional connectivity measured by BOLD signal fluctuations. During this sequence, the participants are asked to fix a white cross on a black background for 8 minutes and leave their thoughts wander. Simultaneous recording of physiological parameters (heart rate and respiration) are employed to account for possible artifacts. (Parameters: 200 blood-oxygenation-level-dependent (BOLD) images with TR = 2400 ms, TE = 30 ms, 38 axial slices, slice thickness = 3.2 mm, flip angle = 85°, acquisition matrix = 94 × 128, field of view = 96 × 128).
MRI Resting State | MRI resting state one week after treatment
  Functional MRI sequence without stimulation (resting-state fMRI) scans are employed to assess the longitudinal changes in regional activity and functional connectivity measured by BOLD signal fluctuations. During this sequence, the participants are asked to fix a white cross on a black background for 8 minutes and leave their thoughts wander. Simultaneous recording of physiological parameters (heart rate and respiration) are employed to account for possible artifacts. (Parameters: 200 blood-oxygenation-level-dependent (BOLD) images with TR = 2400 ms, TE = 30 ms, 38 axial slices, slice thickness = 3.2 mm, flip angle = 85°, acquisition matrix = 94 × 128, field of view = 96 × 128).
MRI Resting State | MRI resting state six month after treatment
  Functional MRI sequence without stimulation (resting-state fMRI) scans are employed to assess the longitudinal changes in regional activity and functional connectivity measured by BOLD signal fluctuations. During this sequence, the participants are asked to fix a white cross on a black background for 8 minutes and leave their thoughts wander. Simultaneous recording of physiological parameters (heart rate and respiration) are employed to account for possible artifacts. (Parameters: 200 blood-oxygenation-level-dependent (BOLD) images with TR = 2400 ms, TE = 30 ms, 38 axial slices, slice thickness = 3.2 mm, flip angle = 85°, acquisition matrix = 94 × 128, field of view = 96 × 128).
MRI Diffusion weighted images | MRI DSI pre-treatment
  Diffusion weighted images (DWI) are acquired to examine the longitudinal changes in white matter integrity and to quantify changes in tracts connecting a priori defined regions of interest. The patient would be warned about a slightly louder sequence sound and will be asked to watch their preferred video or closes their eyes and relax during this last sequence.
  DSI parameters are number of directions = 137, b = 3000 s/mm2, TR = 5100 ms, TE = 80 ms, Voxel size= 1.6x1.6x1.6, field of view = 23.9 cm, 64 axial slices, slice thickness = 1.6 mm.
MRI Diffusion weighted images | MRI DSI one week after treatment
  Diffusion weighted images (DWI) are acquired to examine the longitudinal changes in white matter integrity and to quantify changes in tracts connecting a priori defined regions of interest. The patient would be warned about a slightly louder sequence sound and will be asked to watch their preferred video or closes their eyes and relax during this last sequence.
  DSI parameters are number of directions = 137, b = 3000 s/mm2, TR = 5100 ms, TE = 80 ms, Voxel size= 1.6x1.6x1.6, field of view = 23.9 cm, 64 axial slices, slice thickness = 1.6 mm.
MRI Diffusion weighted images | MRI DSI six month after treatment
  Diffusion weighted images (DWI) are acquired to examine the longitudinal changes in white matter integrity and to quantify changes in tracts connecting a priori defined regions of interest. The patient would be warned about a slightly louder sequence sound and will be asked to watch their preferred video or closes their eyes and relax during this last sequence.
  DSI parameters are number of directions = 137, b = 3000 s/mm2, TR = 5100 ms, TE = 80 ms, Voxel size= 1.6x1.6x1.6, field of view = 23.9 cm, 64 axial slices, slice thickness = 1.6 mm.
Electroencephalography (EEG) resting state | EEG resting state pre-treatment
  All the EEG data are continuously recorded with a sampling rate of 1000 Hz using a 256-electrode Hydrocel cap referenced to the vertex (Cz). Resting-state data with closed eyes is acquired for 6 minutes.
Electroencephalography (EEG) resting state | EEG resting state one week after treatment
  All the EEG data are continuously recorded with a sampling rate of 1000 Hz using a 256-electrode Hydrocel cap referenced to the vertex (Cz). Resting-state data with closed eyes is acquired for 6 minutes.
Electroencephalography (EEG) resting state | EEG resting state six month after treatment
  All the EEG data are continuously recorded with a sampling rate of 1000 Hz using a 256-electrode Hydrocel cap referenced to the vertex (Cz). Resting-state data with closed eyes is acquired for 6 minutes.
EEG auditory | EEG Auditory pre-treatment
  Auditory steady state response paradigm: sequences of 2 types of auditory stimuli are presented binaurally: a 100 ripple tones (40 Hz) and 10 semi-randomly intermixed flat tones (1000 Hz). Ripple tones are presented at about 93 dB and the flat tones at about 83 dB. Participants are asked to detect the flat tone, while the ripple tones entrained the neural gamma oscillatory response. The duration of the task is around 7 minutes.
EEG auditory | EEG Auditory one week after treatment
  Auditory steady state response paradigm: sequences of 2 types of auditory stimuli are presented binaurally: a 100 ripple tones (40 Hz) and 10 semi-randomly intermixed flat tones (1000 Hz). Ripple tones are presented at about 93 dB and the flat tones at about 83 dB. Participants are asked to detect the flat tone, while the ripple tones entrained the neural gamma oscillatory response. The duration of the task is around 7 minutes.
EEG auditory | EEG Auditory six month after treatment
  Auditory steady state response paradigm: sequences of 2 types of auditory stimuli are presented binaurally: a 100 ripple tones (40 Hz) and 10 semi-randomly intermixed flat tones (1000 Hz). Ripple tones are presented at about 93 dB and the flat tones at about 83 dB. Participants are asked to detect the flat tone, while the ripple tones entrained the neural gamma oscillatory response. The duration of the task is around 7 minutes.
EEG visual | EEG Visual pre-treatment
  Visual inward moving grating task paradigm: participants are presented with 3 blocks of 80 trials, with each trial consisting of a circular sinewave grating that contracted toward central fixation. The task of the participants is to detect and respond by button press to a velocity increase of the stimulus, randomly occurring between 750 and 3000 ms. Feedback on performance is provided on every trial, shortly after the response onset terminated stimulus presentation. The duration of the task is around 21 minutes in 3 blocks.
EEG visual | EEG Visual one week after treatment
  Visual inward moving grating task paradigm: participants are presented with 3 blocks of 80 trials, with each trial consisting of a circular sinewave grating that contracted toward central fixation. The task of the participants is to detect and respond by button press to a velocity increase of the stimulus, randomly occurring between 750 and 3000 ms. Feedback on performance is provided on every trial, shortly after the response onset terminated stimulus presentation. The duration of the task is around 21 minutes in 3 blocks.
EEG visual | EEG Visual six month after treatment
  Visual inward moving grating task paradigm: participants are presented with 3 blocks of 80 trials, with each trial consisting of a circular sinewave grating that contracted toward central fixation. The task of the participants is to detect and respond by button press to a velocity increase of the stimulus, randomly occurring between 750 and 3000 ms. Feedback on performance is provided on every trial, shortly after the response onset terminated stimulus presentation. The duration of the task is around 21 minutes in 3 blocks.

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Function (BRIEF) questionnaire | BRIEF pre-treatment
  Children and Adults version. This questionnaire provides an ecological assessment of EF, with a Global Executive Composite (GEC) score derived from the Behavioral Regulation Index (BRI) and Metacognitive Index (MI). The BRI includes subscales of Inhibition, Shifting, Emotional regulation and only in the adult-form, Self- monitoring. The MI includes subscales of Initiation, Working memory, Planning, Organization and Monitoring. Observations are reported using standardized scores (T-scores)
Behavior Rating Inventory of Executive Function (BRIEF) questionnaire | BRIEF one week after treatment
  Children and Adults version. This questionnaire provides an ecological assessment of EF, with a Global Executive Composite (GEC) score derived from the Behavioral Regulation Index (BRI) and Metacognitive Index (MI). The BRI includes subscales of Inhibition, Shifting, Emotional regulation and only in the adult-form, Self- monitoring. The MI includes subscales of Initiation, Working memory, Planning, Organization and Monitoring. Observations are reported using standardized scores (T-scores)
Behavior Rating Inventory of Executive Function (BRIEF) questionnaire | BRIEF six month after treatment
  Children and Adults version. This questionnaire provides an ecological assessment of EF, with a Global Executive Composite (GEC) score derived from the Behavioral Regulation Index (BRI) and Metacognitive Index (MI). The BRI includes subscales of Inhibition, Shifting, Emotional regulation and only in the adult-form, Self- monitoring. The MI includes subscales of Initiation, Working memory, Planning, Organization and Monitoring. Observations are reported using standardized scores (T-scores)

OTHER OUTCOMES:
Sensory-motor conflict 1 | Synchrony condition pre-treatment
  The task uses a robotic device altering sensorimotor processing in participants and inducing mild to moderate hallucinations (presence hallucinations - PH) and passivity experiences. Participants move with their hand a robotic device placed in front of them. A second robot placed behind them reproduced their movements, thus delivering tactile feedback on their back either synchronously (0ms between the movement and the touch, sync) or asynchronously (delay of 500ms, async). Participants rate the strength of robot-induced PH, passivity experiences that they felt during robot manipulation, and control items. Occurrence and severity of clinical symptoms are assessed.
Sensory-motor conflict 1 | Synchrony condition one week after treatment
  The task uses a robotic device altering sensorimotor processing in participants and inducing mild to moderate hallucinations (presence hallucinations - PH) and passivity experiences. Participants move with their hand a robotic device placed in front of them. A second robot placed behind them reproduced their movements, thus delivering tactile feedback on their back either synchronously (0ms between the movement and the touch, sync) or asynchronously (delay of 500ms, async). Participants rate the strength of robot-induced PH, passivity experiences that they felt during robot manipulation, and control items. Occurrence and severity of clinical symptoms are assessed.
Sensory-motor conflict 1 | Synchrony condition six month after treatment
  The task uses a robotic device altering sensorimotor processing in participants and inducing mild to moderate hallucinations (presence hallucinations - PH) and passivity experiences. Participants move with their hand a robotic device placed in front of them. A second robot placed behind them reproduced their movements, thus delivering tactile feedback on their back either synchronously (0ms between the movement and the touch, sync) or asynchronously (delay of 500ms, async). Participants rate the strength of robot-induced PH, passivity experiences that they felt during robot manipulation, and control items. Occurrence and severity of clinical symptoms are assessed.
Sensory-motor conflict 2 | Asynchrony condition pre-treatment
  The task uses a robotic device altering sensorimotor processing in participants and inducing mild to moderate hallucinations (presence hallucinations - PH) and passivity experiences. Participants move with their hand a robotic device placed in front of them. A second robot placed behind them reproduced their movements, thus delivering tactile feedback on their back either synchronously (0ms between the movement and the touch, sync) or asynchronously (delay of 500ms, async). Participants rate the strength of robot-induced PH, passivity experiences that they felt during robot manipulation, and control items. Occurrence and severity of clinical symptoms are assessed.
Sensory-motor conflict 2 | Asynchrony condition one week after treatment
  The task uses a robotic device altering sensorimotor processing in participants and inducing mild to moderate hallucinations (presence hallucinations - PH) and passivity experiences. Participants move with their hand a robotic device placed in front of them. A second robot placed behind them reproduced their movements, thus delivering tactile feedback on their back either synchronously (0ms between the movement and the touch, sync) or asynchronously (delay of 500ms, async). Participants rate the strength of robot-induced PH, passivity experiences that they felt during robot manipulation, and control items. Occurrence and severity of clinical symptoms are assessed.
Sensory-motor conflict 2 | Asynchrony condition six month after treatment
  The task uses a robotic device altering sensorimotor processing in participants and inducing mild to moderate hallucinations (presence hallucinations - PH) and passivity experiences. Participants move with their hand a robotic device placed in front of them. A second robot placed behind them reproduced their movements, thus delivering tactile feedback on their back either synchronously (0ms between the movement and the touch, sync) or asynchronously (delay of 500ms, async). Participants rate the strength of robot-induced PH, passivity experiences that they felt during robot manipulation, and control items. Occurrence and severity of clinical symptoms are assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Eliez, Professor, Principal Investigator — University of Geneva, faculty of medicine
Locations (1):
- Developmental imaging and psychopathology lab, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Latreche C, Maeder J, Mancini V, Schneider M, Eliez S. Effects of risperidone on psychotic symptoms and cognitive functions in 22q11.2 deletion syndrome: Results from a clinical trial. Front Psychiatry. 2022 Oct 26;13:972420. doi: 10.3389/fpsyt.2022.972420. eCollection 2022. PMID 36386982